CLINICAL TRIAL: NCT00245089
Title: Phase II Trial of VAC2.2/VA Therapy for Low-Risk B Group Patients With Rhabdomyosarcoma
Brief Title: Vincristine, Dactinomycin, and Cyclophosphamide in Treating Patients With Embryonal Rhabdomyosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Rhabdomyosarcoma Study Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: JRSG-UHA-PED03-02; CDR0000450162 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Dactinomycin; Cyclophosphamide; Vincristine

INTERVENTIONS:
Biological: dactinomycin
Drug: cyclophosphamide
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vincristine, dactinomycin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vincristine, dactinomycin, and cyclophosphamide together works in treating patients with embryonal rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival rate in patients with low-risk embryonal rhabdomyosarcoma treated with intensive chemotherapy comprising vincristine, dactinomycin, and cyclophosphamide followed by vincristine and dactinomycin.

OUTLINE: Patients receive vincristine IV, dactinomycin IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients then receive vincristine IV and dactinomycin IV on day 1. Treatment repeats every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of embryonal rhabdomyosarcoma

  * Primary operation for pathological diagnosis within the past 42 days
  * The following variants are eligible:

    * Botryoid
    * Spindle cell
    * Anaplastic
* Meets 1 of the following stage criteria:

  * Stage I, clinical group II (N1)

    * Favorable site
    * Any tumor size
    * Microscopic residual disease
    * Lymph nodes clinically positive
  * Stage I, clinical group III (N1)

    * Favorable site (orbit only)
    * Any tumor size
    * Gross residual disease
    * Lymph nodes clinically positive
  * Stage I, clinical group III (N0, NX, N1)

    * Favorable site (except orbit)
    * Any tumor size
    * Gross residual disease
    * Lymph nodes clinically negative, involvement unknown, or positive
  * Stage II, clinical group II (N0, NX)

    * Unfavorable site
    * Small tumor (≤ 5 cm in diameter)
    * Microscopic residual disease
  * Stage III, clinical group I or II (N0, NX, N1)

    * Unfavorable site
    * Small tumor (≤ 5 cm in diameter) with positive nodes or large tumor (> 5 cm in diameter) with any lymph nodes status
    * Completely resected or microscopic residual disease

PATIENT CHARACTERISTICS:

Performance status

* 0-3

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 7.5 g/dL

Hepatic

* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Bile acid ≤ 2.5 times ULN

Renal

* Creatinine based on age as follows:

  * ≤ 0.8 mg/dL (for patients < 5 years of age)
  * ≤ 1.2 mg/dL (for patients 5-9 years of age)
  * ≤ 1.5 mg/dL (for patients ≥ 10 years of age)

Cardiovascular

* No severe heart disease

Other

* Not pregnant or nursing
* No uncontrolled infection
* Must have acceptable organ function for age
* No other malignancy within the past 5 years
* No hypersensitivity attributed to study drugs
* No Charcot-Marie-Tooth disease or chickenpox

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior anticancer chemotherapy

Endocrine therapy

* Prior anticancer steroids allowed

Radiotherapy

* Prior emergency radiotherapy allowed within the past 2 weeks

Other

* No concurrent pentostatin

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Estimated)
Dates: Start 2004-05; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival at 3 years after study registration

SECONDARY OUTCOMES:
Overall survival at 3 years after study registration
Toxicity by NCI CTC at 3 years after study registration

CONTACTS AND LOCATIONS:
Overall Officials: Hajime Hosoi, Study Chair — Kyoto Prefectural University of Medicine; Ryoji Hanada, MD — Saitama Children's Medical Center; Keizo Horibe, MD, PhD — National Hospital Orgnization Nagoya Medical Center
Locations (48):
- Japan (48):
  - Anjo Kosei Hosptial, Anjo, Aichi-ken
  - Aichi Medical University, Nagakuti, Aichi-ken
  - National Hospital Orgnization Nagoya Medical Center, Nagoya, Aichi-ken
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kurume University School of Medicine, Kurume, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gifu University Graduate School of Medicine, Gifu, Gifu
  - Gunma Children's Medical Center, Seta-gun, Gunma
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization - Medical Center of Kure, Kure, Hiroshima
  - Sapporo Medical University, Sapporo, Hokkaido
  - Hokkaido University Graduate School of Medicine, Sapporo, Hokkaido
  - Kobe City General Hospital, Kobe, Hyōgo
  - Ibaraki Children's Hospital, Mito, Ibaraki
  - University of Tsukuba, Tsukuba, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University, Kanazawa, Ishikawa-ken
  - Kagoshima University, Kagoshima, Kagoshima-ken
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - National Center for Child Health and Development, Tokyo, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Yokohama City University, Yokohama, Kanagawa
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Miyazaki Medical College University of Miyazaki, Miyazaki-gun, Miyazaki
  - Nagano Children's Hospital, Toyoshina-machi, Nagano
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Osaka City University, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka City General Hospital, Suita-shi, Osaka
  - Osaka University Graduate School of Medicine, Suita-shi, Osaka
  - Osaka Medical College, Takatsuki, Osaka
  - Dokkyo University School of Medicine, Koshigaya, Saitama
  - Saitama Children's Medical Center, Saitama, Saitama
  - National Defense Medical College, Tokorozawa, Saitama
  - Shiga University of Medical Science, Ōtsu, Shiga
  - Shimane University Hospital, Izumo, Shimane
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - National Cancer Center Hospital, Tokyo, Tokyo
  - St. Luke's International Hospital, Tokyo, Tokyo
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - Toho University School of Medicine, Tokyo, Tokyo
  - Keio University School of Medicine, Tokyo, Tokyo
  - Nihon University Itabashi Hospital, Tokyo, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Hokkaido Medical Center for Child Health and Rehabilitation, Sapporo